CLINICAL TRIAL: NCT01302132
Title: An Open Label Study to Evaluate the Pharmacokinetics of ASP1941 After a Single Oral Dose of 14C-labeled ASP1941 in Healthy Male Subjects
Brief Title: Mass Balance Study of ASP1941
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1941-CL-0055; 2008-000316-33 (EudraCT Number)
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects
Keywords: Mass Balance; ASP1941; Pharmacokinetics
MeSH Terms: interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ASP1941 — Oral solution

SUMMARY:
This study investigates the pharmacokinetics, in particular the routes and extent of metabolism and excretion, of ASP1941 after a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 60-100kg, BMI between 18.5-30 kg/m2, inclusive

Exclusion Criteria:

* Pulse <40 or >90 bpm; Systolic Blood Pressure > 140 mmHg; Diastolic Blood Pressure >90 mmHg

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP1941 to evaluate metabolism and excretion | up to 216 hours

SECONDARY OUTCOMES:
Identification of metabolic profile of ASP1941 | up to 216 hours

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Zuidlaren, Netherlands